CLINICAL TRIAL: NCT02535013
Title: Benefit of Intraoperative Lung Ultrasound in Pediatric Patients Undergoing Cardiac Surgery
Brief Title: Intraoperative Lung Ultrasound in Pediatric Patients
Acronym: LUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1507-062-687
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Ultrasonography; Pediatrics; Perioperative Period; Lung; Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): No intervention during the perioperative period. Perform lung ultrasound twice only for the diagnostic purpose at the end of surgery and 6 to 12 hours after surgery in the intensive care unit.
  Interventions: Device: Lung ultrasound
- Ultrasound (Active Comparator): Perform lung ultrasound three times during the perioperative period; after the induction of general anesthesia, at the end of surgery, and 6 to 12 hours after surgery in the intensive care unit. According to the lung ultrasound finding, conduct appropriate interventions such as, alveolar recruitment maneuver for atelectasis, or chest tube insertion for pneumothorax.
  Interventions: Device: Lung ultrasound

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasound with appropriate interventions depending on the ultrasound finding

SUMMARY:
Investigators hypothesized that perioperative lung ultrasound would be beneficial in pediatric patients undergoing cardiac surgery compared to those who did not receive lung ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Acyanotic congenital heart disease patients undergoing cardiac surgery under general anesthesia

Exclusion Criteria:

* History of surgery on the lungs
* Cyanotic congenital heart disease
* Abnormal preoperative chest radiograph findings including atelectasis, pneumothorax, pleural effusion, and pneumonia
* Considered inappropriate by the investigator

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Intraoperative incidence of pulse oximetry (SpO2) ≤ 95% (or 10% below the baseline value) | from the induction of general anesthesia until the end of the surgery, up to 24 hours
Postoperative incidence of SpO2 ≤ 95% (or 10% below the baseline value) | within the first day after surgery
Postoperative incidence of respiratory complications | within the first day after surgery

SECONDARY OUTCOMES:
Intraoperative partial pressure of oxygen in arterial blood (PaO2) from arterial blood gas analysis | from the induction of general anesthesia until the end of the surgery, up to 24 hours
Postoperative partial pressure of oxygen in arterial blood (PaO2) from arterial blood gas analysis | within the first day after surgery
Initial SpO2 on arriving at pediatric intensive care unit | from the end of the surgery until postoperative 1 hour
Days needed to wean from mechanical ventilation | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lutterbey G, Wattjes MP, Doerr D, Fischer NJ, Gieseke J Jr, Schild HH. Atelectasis in children undergoing either propofol infusion or positive pressure ventilation anesthesia for magnetic resonance imaging. Paediatr Anaesth. 2007 Feb;17(2):121-5. doi: 10.1111/j.1460-9592.2006.02045.x. PMID 17238882
- [Background] Tusman G, Bohm SH, Tempra A, Melkun F, Garcia E, Turchetto E, Mulder PG, Lachmann B. Effects of recruitment maneuver on atelectasis in anesthetized children. Anesthesiology. 2003 Jan;98(1):14-22. doi: 10.1097/00000542-200301000-00006. PMID 12502973
- [Background] Bronicki RA, Chang AC. Management of the postoperative pediatric cardiac surgical patient. Crit Care Med. 2011 Aug;39(8):1974-84. doi: 10.1097/CCM.0b013e31821b82a6. PMID 21768801
- [Background] Vitale V, Ricci Z, Cogo P. Lung ultrasonography and pediatric cardiac surgery: first experience with a new tool for postoperative lung complications. Ann Thorac Surg. 2014 Apr;97(4):e121-4. doi: 10.1016/j.athoracsur.2014.01.060. PMID 24694455
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376